CLINICAL TRIAL: NCT07192731
Title: Treatment of LIVER-limited HepatoCellular Carcinoma (HCC) in Patients With Preserved Liver Function by IRreversible Electroporation: A Prospective, International, Multi-centre Cohort Study
Brief Title: International Study on Treatment of Liver (HCC) Patients With IRE
Acronym: LIVERHCC-IRE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Angiodynamics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-ONC-02
Record Dates: First submitted 2025-09-23; First posted 2025-09-25 (Actual); Last update posted 2025-10-10 (Actual); Status verified 2025-10

CONDITIONS: Hepatocellular Carcinoma (HCC); Liver Ablation; Liver Cancer, Adult
Keywords: irreversible electroporation; liver ablation; nanoknife; liver ire registry
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Electroporation

STUDY DESIGN:
Intervention Model Description: This is an international, prospective, multi-centre, registry-based, non-randomized, single arm clinical cohort study of the use of IRE for the treatment of HCC
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Other: Use of NanoKnife System for ablation of HCC lesions (Experimental)
  Interventions: Device: Irreversible Electroporation

INTERVENTIONS:
Device: Irreversible Electroporation — Irreversible electroporation (IRE) is a procedure which involves the passage of short intense electrical pulses between probes to destabilize cell membranes by creating "nanopores" which leads to cell destabilisation and cell death.
  IRE can be used to selectively damage cancerous cells whilst sparing adjacent supporting connective tissue in vessels and bile ducts allowing a more targeted treatment compared to other types of ablation. IRE also avoids the heat-sink phenomenon which compromises the effectiveness of thermal ablation and possibly reduces the risks of biliary injury.
  Other Names: nanoknife

SUMMARY:
Procedural data will be recorded from patients with liver lesions from hepatocellular cancer who have been assessed by an appropriately constituted MDT (or equivalent) as appropriate to receive irreversible electroporation

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years and over, able to provide informed consent and with clinical diagnosis of an HCC. Tissue confirmation of HCC prior to treatment is not standard of care and is therefore not required for this study.
* Child-Pugh A up to A6.
* Eastern Co-operative Oncology Group (ECOG) Score ≤ 2.
* Rockwood Frailty Score ≤ 3.
* Serum bilirubin < 30 µmol/L.
* Serum creatinine < 150 µmol/L.
* No extrahepatic metastases
* IRE can be used for up to 3 tumours < 3cm in size. Other forms of ablation can be combined with IRE in the same sitting but not for the same lesion. IRE can also be combined with surgical resection.

Exclusion Criteria:

General:

* Patients involved in other research studies.
* Patients under the age of 18 years.
* Inability to give informed consent.
* Patients who are pregnant.
* Child-Pugh B or C.
* Patients with an ECOG status of > 2 at time of recruitment.
* Rockwood Frailty Score > 3
* Impaired renal function (serum creatinine > 150 µmol/L)
* Accepted exclusions to IRE from consensus criteria including:
* Platelet count < 50x109 U/L.
* International normalised ratio (INR) for blood clotting > 1.7.
* Prior hepatic tumour ablation.

Cardiovascular fitness related exclusions:

* History of ventricular arrhythmia.
* Implanted pacemaker or defibrillator.
* Congestive cardiac failure NYHA Class ≥ 3.

Tumour-related exclusions:

* Tumour ≥ 3 cm in size.
* Extrahepatic metastatic disease.
* Jaundice (serum bilirubin > 30 µmol/L).
* MDT recommends use of thermal ablation for any given lesion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2028-02 (Estimated); Study Completion 2029-02 (Estimated)

PRIMARY OUTCOMES:
Target Tumour Eradication | 6 months
  The percentage of target tumours successfully eradicated 6 months after the initial IRE procedure, according to RECIST and PERCIST criteria. This is based on a per-lesion analysis.

SECONDARY OUTCOMES:
Complications of IRE: Episode-related complications: | 30 days
  Episode-related complications of IRE using the Clavien-Dindo system and the comprehensive complication index (CCI)
Complications of IRE: Intervention for local liver-related complications of IRE | 12 months
  Any intervention for local liver-related complications of IRE within 12 months of procedure. Interventions will be categorised as radiological, surgical or medical.
Oncological outcomes: Incomplete ablation requiring further intervention | 6 months
  Re-ablation and modality.
Oncological Outcome: Progression at site of ablation | 12 months
  Appearance of new lesions in liver, lungs, peritoneum or elsewhere (other) on follow-up.
Oncological outcome: Further anti-cancer intervention | 12 months
  Any further liver-directed, anti-cancer intervention including TACE and SIRT
Oncological Outcome: Survival (Progression-free & overall) | 12 months
  Progression-free and overall survival at 12 months from time of IRE.
Oncologic Outcomes: local progression | 12 months
  Local progression at site of IRE-treated lesion.
Oncologic Outcomes: Chemotherapy post-IRE | 6 months
  Any use of chemotherapy after IRE.
Quality of life: EQ-5D-5 pre-procedure | within 7 days prior to procedure
  Effect of intervention on quality of life as assessed by EQ-5D-5
Quality of life: EQ-5D-5 post-procedure 7 days | 7 days
  Effect of intervention on quality of life as assessed by EQ-5D-5
Quality of life: EQ-5D-5 - 6 months | 6 months
  Effect of intervention on quality of life as assessed by EQ-5D-5

CONTACTS AND LOCATIONS:
Overall Officials: Ajith Siriwardena, MD FRCS, Principal Investigator — Manchester Royal Infirmiary
Locations (1):
- Manchester Royal Infirmiary, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided